CLINICAL TRIAL: NCT05765422
Title: Sport and Health a Pilot Study: Impact of Endurance Physical Activity on the Microbiological Homeostasis of the Oral Cavity of Young Adults
Brief Title: The Influence of Endurance Sports Activity on the Oral Microbiota of Young Adults.
Acronym: ORAMICAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22-PP-11
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sedentary (Other): Participant does not meet WHO's recommendations with the physical activity
  Interventions: Other: salivar and gum sampling
- OMS recommandations (Other): Participant does not meet WHO's recommendations (2.5-5 hours per week of moderate physical activity OR 1.25-2.5 hours per week of vigorous physical activity);
  Interventions: Other: salivar and gum sampling
- More than the OMS recommandations (Other): Participant is practicing physical activity more than the WHO recommendations
  Interventions: Other: salivar and gum sampling

INTERVENTIONS:
Other: salivar and gum sampling — Saliva will then be collected by salivary spit and a mucosal smear will be taken using a swab passed at the junction of the tooth and the gum

SUMMARY:
The oral cavity is an easily accessible anatomical site that accurately reflects the health of the individual. The mouth is considered an early indicator of biological aging, leading to the identification of oral biomarkers predictive of future alterations. Current data show that the oral health of high level athletes is globally altered with an increase in cariogenic indexes, an increased incidence of periodontitis, dental trauma and dry mouth syndromes. Few studies have focused on the oral microbiota compared to mouthguards used in rugby or boxing which seem to induce dysbiosis, a recent study shows an effect of ketogenic diet on bacterial changes in the mouth of endurance athletes. This project focuses on the impact of intensive sport practice on oral health and the identification of oral biomarkers associated with physical activity. The objective of this study is to investigate the impact of the amount of endurance sport practice on oral microbiota and oral health in young adults. the hypothesis is that a sedentary lifestyle and high-level sport induce depletion and/or changes in the oral microbiota compared to regular physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 30 years old
* If practicing sports, it must be an endurance sport as main activity (cycling or running)

Exclusion Criteria:

* Practice more than 3 hours of swimming per week
* Have taken anti-inflammatory drugs, less than 48 hours before the study
* Have taken antibiotics and/or probiotics, less than 3 weeks before the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Analysis of the oral microbiota in healthy individuals engaged in endurance physical activity at different levels. | 3 years
  Microbiological screening will be performed using an innovative methodology based on microfluidic PCR (BiomarkHD) (number of bacterial colonies)

SECONDARY OUTCOMES:
Quantification of salivary inflammatory markers in healthy individuals who perform endurance physical activity at different levels. | 3 years
  numer and type of salivary inflammatory markers will performed using multiplex analysis technology developed by the firm Meso Scale Diagnostic (MSD).

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ortis M, Dubois M, Bougault V, Legueult K, Fassy J, Mari B, Bertrand MF, Lupi L, Doglio A. ORASPORT study protocol: a prospective observational study on the impact of endurance physical activity on oral microbiology and immunology. Front Oral Health. 2025 Dec 5;6:1692359. doi: 10.3389/froh.2025.1692359. eCollection 2025. PMID 41424657